CLINICAL TRIAL: NCT05260554
Title: Effects of Use of Cranberry Extract Instead of Antibiotics During Uncomplicated Urinary Tract Infection
Brief Title: Effect of Cranberry Extract on the Urinary System
Status: Completed | Type: Observational
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Oya Guven, MD, Assistant Professor, Kırklareli University
Other Study IDs: Kırklareli University
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Urinary Tract Disease; Cystitis; Antibiotic Reaction
Keywords: Urinary Tract Disease; Cranberry extract; Antibiotic; Cystitis
MeSH Terms: conditions — Urologic Diseases; Cystitis | interventions — Fosfomycin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- using fosfomycin: The patients in this group; have been prescribed fosfomycin for 7 days (3 doses, two days apart).
  Interventions: Drug: Fosfomycin
- using cranberry extract: The patients in this group; took 7 days (1 tablet each day) of cranberry tablets.
  Interventions: Dietary Supplement: Cranberry

INTERVENTIONS:
Drug: Fosfomycin — In this group with urinary tract inflammation; Fosfomycin was prescribed for 7 days (3 doses, 2 days apart). There are 80 patients in total.
  Other Names: monurol
  Groups: using fosfomycin
Dietary Supplement: Cranberry — In this group with urinary tract inflammation; 7 days (used every day) cranberry tablet was given. There are 80 patients in total.
  Groups: using cranberry extract

SUMMARY:
In this study, we will try to emphasize the effects of using cranberry tablets, which is an alternative to antibiotic therapy, during uncomplicated urinary tract infections (only urinary tract, bladder and kidney infections did not).

DETAILED DESCRIPTION:
This study was Istanbul Kartal Dr. Lütfi Kırdar Training and Research Hospital Emergency Medicine Clinic and Kırklareli Training and Research Hospital Emergency Service and Internal Medicine Polyclinic. Our study; includes patients who applied to the Emergency Department and Internal Medicine outpatient clinic with the complaint of dysuria and had normal WBC, CRP, urea, and creatinine values in their analysis, and leukocyturia was found in the urine test. Two options were offered in the treatment to these patients. Vaccinium Macrocarpon Aiton preparation or fosfomycin was given for seven days. The patients were asked whether their complaints had decreased according to the Lykert-Type verbal scale at the time of admission and on the first, third, and seventh days. When the treatment was finished, leukocytes were checked in the urinalysis. This outcome was compared between the 2 treatment options. We also noted whether nausea.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18
* who have urinary tract inflammation
* who haven't kidney dissease previous

Exclusion Criteria:

* Younger than 18
* Who have kidney inflammation
* Pregnant patients
* Who have blood test abnormal (WBC, Ure, Creatin, CRP high level)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among the patients who were eligible criteria, the study was terminated when the number of patients in both groups reached 80.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Treatment time | 7 days
  After 7 days of treatment, the 2 treatment options were compared with each other.

CONTACTS AND LOCATIONS:
Overall Officials: Oya Guven, Study Director — Kırklareli University
Locations (1):
- Oya Guven, MD, Kırklareli, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data results of the patients will be described in the article.

REFERENCES:
- [Result] Gray M. Are cranberry juice or cranberry products effective in the prevention or management of urinary tract infection? J Wound Ostomy Continence Nurs. 2002 May;29(3):122-6. doi: 10.1067/mjw.2002.124016. No abstract available. PMID 12011903